CLINICAL TRIAL: NCT06801197
Title: Impact of a Mobile App-Based Waitlist Intervention (MI-Coach: ED) on Readiness for Eating Disorder Treatment: a Randomized Controlled Trial
Brief Title: Impact of a Mobile App-Based Waitlist Intervention on Readiness for Eating Disorder Treatment
Acronym: MI-Coach: ED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Maya Libben, Associate Professor of Psychology, University of British Columbia
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: H24-03392; 24901 (Other Grant/Funding Number: Social Sciences and Humanities Research Council (SSHRC))
Record Dates: First submitted 2025-01-21; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Eating Disorders
Keywords: eating disorders; digital interventions; motivational interviewing; treatment barriers
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: The study employs a sequential interventional study design to evaluate the MI-Coach: ED app, ensuring both ethical considerations and robust data collection. Participants are randomized into two groups: the treatment group, which uses the app immediately for four weeks, and the delayed treatment control group, which remains on the waitlist without intervention for four weeks before gaining access to the app. Both groups complete weekly motivation assessments and pre- and post-intervention questionnaires at 0, 4, 8, and 12 weeks. This design allows for between-group comparisons during the initial phase and within-group comparisons after the delayed group transitions to the intervention, capturing immediate, delayed, and sustained effects of the app. By reflecting real-world waitlist scenarios, this model ensures all participants benefit from the intervention while providing valuable longitudinal data to assess its efficacy and practical application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Immediate Treatment Group (MI-Coach: ED Users) (Experimental): Participants randomized to the immediate treatment group will begin using the MI-Coach: ED app immediately for a four-week intervention period. During this time, participants will complete interactive modules designed to enhance motivation and readiness for treatment, focusing on topics such as ambivalence, self-acceptance, compassionate motivation, and behavior change strategies. Weekly brief assessments of motivation and readiness for change will be completed throughout the initial four-week period.
  Interventions: Combination Product: MI-Coach: ED Mobile App
- Delayed Treatment Group (Waitlist Control) (No Intervention): Participants randomized to the delayed treatment group will remain on the waitlist without access to the MI-Coach: ED app for the first four weeks. During this period, participants will complete weekly brief assessments of motivation and readiness for change to evaluate changes while waiting for access to the intervention. No additional interventions or activities will be provided during this initial four-week period.
- Combined Treatment Group (Experimental): This arm includes all participants who engage with the MI-Coach: ED app during the eight weeks following the initial four-week period. Participants from the immediate treatment group (Arm 1) will continue to use the app for the full 12 weeks of the study, including an eight-week extended intervention period and follow-up assessments at 8 and 12 weeks to evaluate the app's sustained effects. Participants transitioning from the delayed treatment group (Arm 2) will also use the app for an eight-week intervention period after their initial four-week waitlist phase, ensuring both groups have the same opportunity to complete the full intervention. Weekly assessments of motivation and readiness for change will continue for all participants during their respective intervention periods, along with follow-up assessments to compare immediate and delayed access effects, as well as the app's long-term impact on motivation and clinical outcomes.
  Interventions: Combination Product: MI-Coach: ED Mobile App

INTERVENTIONS:
Combination Product: MI-Coach: ED Mobile App — The MI-Coach: ED mobile app is a self-guided intervention designed to enhance motivation and readiness for treatment in adults with eating disorders. The app includes seven sequential modules based on motivational interviewing (MI) principles, addressing ambivalence, self-acceptance, compassionate motivation, behavior change goals, sustain and change talk, commitment language, and relapse prevention. Each module incorporates interactive content, including educational videos, articles, and exercises, tailored to support motivation across a range of eating disorder diagnoses. The app is designed to be user-friendly and scalable, providing an accessible, cost-effective solution for individuals on waitlists for formal eating disorder treatment.
  Arms: Combined Treatment Group; Immediate Treatment Group (MI-Coach: ED Users)

SUMMARY:
The goal of this randomized controlled trial is to evaluate whether a mobile app-based motivational interviewing intervention (MI-Coach: ED) can improve motivation and readiness for treatment in adults with eating disorders who are currently on waitlists for provincially funded eating disorder services in British Columbia. The main questions it aims to answer are:

* Does the use of MI-Coach: ED improve overall motivation, confidence, and readiness for treatment compared to treatment-as-usual (waitlist with no intervention)?
* Does the app help mitigate declines in motivation over time among waitlisted individuals?

Researchers will compare participants using the MI-Coach: ED app to a delayed treatment control group to assess differences in motivation, readiness for treatment, and associated clinical outcomes.

Participants will:

* Treatment group: Use the MI-Coach: ED app for four weeks, completing interactive modules focused on motivation and readiness for change, while also completing weekly brief assessments of motivation.
* Delayed treatment group: Remain on the waitlist with no intervention for four weeks while completing weekly brief assessments of motivation. After this period, they will receive access to the MI-Coach: ED app and be integrated into the treatment group.
* Complete pre-test and post-test questionnaires at 0, 4, 8, and 12 weeks assessing motivation, eating pathology, anxiety, and depressive symptoms.

This study aims to inform evidence-based practices for reducing the adverse effects of long waitlist durations on individuals with eating disorders.

DETAILED DESCRIPTION:
This study is a randomized controlled trial designed to evaluate the efficacy of MI-Coach: ED, a mobile app-based intervention tailored for adults with eating disorders (EDs) currently on waitlists for provincially funded ED treatment programs in British Columbia, Canada. The study explores how a scalable, self-guided digital tool can support motivation and readiness for treatment during a critical period when access to traditional care is delayed.

MI-Coach: ED leverages evidence-based principles of motivational interviewing (MI) to address ambivalence and enhance intrinsic motivation to engage in treatment. The app features seven interactive modules covering key topics, including self-acceptance, behavior change strategies, and relapse prevention, delivered through videos, exercises, and self-reflection activities. These modules aim to foster readiness for treatment, improve confidence, and maintain motivation during extended wait times.

The trial uses a sequential interventional study design. Participants are randomized into two groups: a treatment group that begins using the MI-Coach: ED app immediately for four weeks and a delayed treatment control group that waits four weeks before accessing the intervention. Both groups complete regular assessments of motivation, readiness for change, eating pathology, anxiety, depressive symptoms, and other clinical characteristics at baseline, 4 weeks, 8 weeks, and 12 weeks. In-app engagement metrics, such as module completion rates, are also collected to evaluate feasibility and acceptability.

This trial incorporates exploratory analyses to investigate the impact of app use on broader clinical outcomes, such as body dissatisfaction and mental health symptoms, and examines whether app engagement predicts clinical improvements. Statistical methods include descriptive analyses, t-tests for between-group comparisons, and linear mixed modeling (LMM) to evaluate longitudinal changes.

The findings aim to inform the integration of digital tools into clinical practice, offering evidence for their utility in mitigating the adverse effects of waitlist delays. By addressing a critical gap in care for individuals with EDs, this study seeks to enhance the accessibility and effectiveness of pre-treatment interventions and contribute to the development of more comprehensive care pathways.

ELIGIBILITY:
Inclusion Criteria:

* Must self-identify as a woman, including cisgender or transgender individuals.
* Must be at least 18 years old at the time of enrollment.
* Currently on a waitlist to receive treatment for an eating disorder at provincially funded eating disorder programs in British Columbia.
* Meets criteria for a threshold or subthreshold eating disorder, including anorexia nervosa (restricting or binge/purge subtype), bulimia nervosa, binge eating disorder, or other specified feeding or eating disorder (OSFED).
* Able to read and understand English fluently.
* Owns or has regular access to a smartphone or mobile device capable of running the MI-Coach: ED app.

Exclusion Criteria:

* Does not identify as a woman, regardless of sex assigned at birth.
* Currently receiving active treatment for an eating disorder, such as outpatient therapy, inpatient care, or day programs.
* Diagnosed with a schizophrenia-spectrum disorder or other psychotic disorder.
* Presence of a cognitive impairment or sensory deficit (e.g., severe visual or hearing impairment) that would interfere with the ability to use the app or complete study assessments.
* History of a recent traumatic brain injury or neurological condition that might impact participation.
* Any condition that, in the opinion of the investigators, would interfere with the participant's ability to comply with the study protocol or complete the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is open to individuals who self-identify as women, including cisgender women and transgender individuals who identify as women. The inclusion criteria are based on self-reported gender identity, ensuring the study captures the experiences of a diverse group of women. Individuals who do not identify as women, regardless of sex assigned at birth, are not eligible to participate in this trial. This criterion is intended to align with the study's focus on evaluating the MI-Coach: ED app within this specific population.
Enrollment: 74 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Overall Motivation for Treatment as Measured by the Readiness and Motivation Questionnaire (RMQ) at 4 Weeks | From enrollment to the end of initial study arm at 4 weeks
  Overall motivation for treatment will be assessed using the Readiness and Motivation Questionnaire (RMQ), a validated measure evaluating readiness to change eating disorder symptoms and behaviors. The RMQ provides a total motivation score (ranging from 0 to 100) and includes subscales for precontemplation, action, internality, and confidence. Higher scores indicate greater readiness for treatment. Changes from baseline to 4 weeks will be evaluated using linear mixed modeling (LMM), accounting for fixed effects (treatment group, time) and random effects (individual variability). A significant change from baseline will be defined as a statistically significant fixed effect of time (p < 0.05), with a greater increase in motivation scores observed in the treatment group compared to the delayed treatment control group.
Rate of Change in Weekly Motivation Levels as Measured by the Motivational Stages of Change for Adolescents Recovering from an Eating Disorder (MSCARED) During the Initial 4 Weeks | From enrollment to the end of initial study arm at 4 weeks
  Weekly motivation will be assessed using the Motivational Stages of Change for Adolescents Recovering from an Eating Disorder (MSCARED), a single-item self-report measure. Participants select their current stage of change from six stages: precontemplation, contemplation, preparation, action, maintenance, and recovery. Rate of change will be calculated using LMM, incorporating interaction terms between treatment group and time to evaluate differences in the trajectory of weekly motivation. A significant result will be defined as a statistically significant interaction term (p < 0.05), indicating a slower decline or greater increase in motivation over time in the treatment group compared to the delayed treatment control group.
Change from Baseline in Confidence to Engage in Treatment as Measured by the Confidence Subscale of the Readiness and Motivation Questionnaire (RMQ) at 4 Weeks | From enrollment to the end of initial study arm at 4 weeks
  Confidence to engage in treatment will be assessed using the confidence subscale of the RMQ, which measures participants' belief in their ability to address eating disorder behaviors. Scores range from 0 to 100, with higher scores indicating greater confidence. Changes from baseline to 4 weeks will be analyzed using LMM, incorporating fixed effects for treatment group and time, and random effects for individual differences. A significant change from baseline will be defined as a statistically significant fixed effect of time (p < 0.05), with confidence scores in the treatment group showing stability or improvement compared to the delayed treatment control group.

SECONDARY OUTCOMES:
Attrition Rate Between Baseline and 4 Weeks | From enrollment to the end of initial study arm at 4 weeks
  Attrition will be measured as the percentage of participants who do not complete study activities (e.g., assessments or app usage) within the first 4 weeks. Descriptive statistics, including means, percentages, and ranges, will be calculated to summarize attrition rates for both groups. Simple t-tests will be used to compare mean attrition rates between the treatment and delayed treatment control groups, with a significant difference defined as a p-value < 0.05, indicating lower attrition in the treatment group.
Participant Ratings of App Acceptability as Measured by the User Version of the Mobile App Rating Scale (uMARS) | At 12 weeks
  Acceptability of the MI-Coach: ED app will be assessed using the User Version of the Mobile App Rating Scale (uMARS). This scale includes subscales for engagement, functionality, aesthetics, and information quality, each rated on a 5-point Likert scale (1 = inadequate, 5 = excellent). Descriptive statistics (means, standard deviations, ranges) will summarize acceptability scores for each subscale and overall scores. Scores averaging ≥ 4 will indicate a "high" or "very high" level of acceptability for the app.
Association Between App Usability and Module Completion Rates | At 12 weeks
  App usability will be assessed using the ease of use and perceived usefulness subscales of the uMARS. Engagement metrics, including the number of modules completed, days the app was used, assessments and exercises completed, and logins, will be obtained from in-app data provided by Resiliens Inc. Generalized linear regression models will evaluate the relationship between usability scores and app engagement metrics, with significant associations defined as a p-value < 0.05. Descriptive statistics will summarize app engagement metrics.

OTHER OUTCOMES:
Exploratory Analysis of Changes in Anxiety Symptoms as Measured by the Generalized Anxiety Disorder-7 (GAD-7) Scale | Baseline, 4 weeks, and follow-ups at 8 and 12 weeks
  Anxiety symptoms will be assessed using the GAD-7, a validated self-report measure with scores ranging from 0 to 21 (higher scores indicate greater severity of anxiety symptoms). Descriptive statistics, including means and standard deviations, will summarize anxiety scores at baseline, 4 weeks, and follow-up time points. Exploratory analyses will use simple t-tests to compare changes in mean anxiety scores between the treatment and delayed treatment control groups at 4 weeks. Changes over time will also be analyzed using linear mixed modeling (LMM) to evaluate group differences in trajectories. Statistical significance will be defined as p < 0.05 for group comparisons or time effects.
Exploratory Analysis of Changes in Body Dissatisfaction as Measured by the Body Shape Questionnaire (BSQ) | Baseline, 4 weeks, and follow-ups at 8 and 12 weeks
  Body dissatisfaction will be assessed using the BSQ, a 34-item self-report measure with scores ranging from 34 to 204 (higher scores indicate greater dissatisfaction with body shape). Descriptive statistics will summarize scores at baseline, 4 weeks, and follow-up time points. Simple t-tests will compare mean changes in body dissatisfaction scores between the treatment and delayed treatment control groups at 4 weeks. LMM will explore whether group differences emerge in body dissatisfaction trajectories across time points, with statistical significance defined as p < 0.05.
Exploratory Analysis of App Engagement Metrics and Clinical Outcomes | Baseline, 4 weeks, and follow-ups at 8 and 12 weeks
  App engagement metrics, including the number of modules completed, days the app was used, assessments and exercises completed, and logins, will be extracted from in-app data provided by Resiliens Inc. Exploratory analyses will examine associations between engagement metrics and changes in clinical outcomes (e.g., motivation, anxiety, body dissatisfaction). Generalized linear regression models will evaluate the predictive relationship between engagement metrics (independent variables) and changes in outcome measures (dependent variables). Descriptive statistics will summarize engagement patterns, and statistical significance will be defined as p < 0.05 for predictive associations.
Exploratory Analysis of Changes in Eating Disorder Symptomatology Over Time | Baseline, 4 weeks, and follow-ups at 8 and 12 weeks
  Eating disorder symptomatology will be assessed using the RMQ symptom-specific subscales (e.g., cognitive, bingeing, compensatory strategies, restriction), with scores ranging from 0 to 100. Exploratory analyses will examine changes in symptom-specific subscale scores between the treatment and delayed treatment control groups using t-tests for between-group differences at 4 weeks and LMM to evaluate changes over time. Descriptive statistics will summarize baseline and follow-up scores, with statistical significance defined as p < 0.05 for group differences or time effects.
Exploratory Analysis of Changes in Depressive Symptoms as Measured by the Patient Health Questionnaire-9 (PHQ-9) Over Time | Baseline, 4 weeks, and follow-ups at 8 and 12 weeks
  Depressive symptoms will be assessed using the PHQ-9, with scores ranging from 0 to 27 (higher scores indicate greater depressive severity). Exploratory analyses will compare changes in PHQ-9 scores between the treatment and delayed treatment control groups at 4 weeks using t-tests. LMM will analyze trajectories over time to explore whether differences emerge between groups. Descriptive statistics will summarize scores at baseline and follow-ups, with significance defined as p < 0.05.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weiss CV, Mills JS, Westra HA, Carter JC. A preliminary study of motivational interviewing as a prelude to intensive treatment for an eating disorder. J Eat Disord. 2013 Aug 20;1:34. doi: 10.1186/2050-2974-1-34. eCollection 2013. PMID 24999413
- [Background] Linardon J, Shatte A, Messer M, Firth J, Fuller-Tyszkiewicz M. E-mental health interventions for the treatment and prevention of eating disorders: An updated systematic review and meta-analysis. J Consult Clin Psychol. 2020 Nov;88(11):994-1007. doi: 10.1037/ccp0000575. Epub 2020 Aug 27. PMID 32852971
- [Background] Keegan E, Waller G, Tchanturia K, Wade TD. The potential value of brief waitlist interventions in enhancing treatment retention and outcomes: a randomised controlled trial. Cogn Behav Ther. 2024 Nov;53(6):608-620. doi: 10.1080/16506073.2024.2351867. Epub 2024 May 9. PMID 38721888
- [Background] Iyar MM, Cox DW, Kealy D, Srikameswaran S, Geller J. Is stage of change enough? Confidence as a predictor of outcome in inpatient treatment for eating disorders. Int J Eat Disord. 2019 Mar;52(3):283-291. doi: 10.1002/eat.23026. Epub 2019 Jan 30. PMID 30701590
- [Background] Innes NT, Clough BA, Casey LM. Assessing treatment barriers in eating disorders: A systematic review. Eat Disord. 2017 Jan-Feb;25(1):1-21. doi: 10.1080/10640266.2016.1207455. Epub 2016 Aug 2. PMID 27485375
- [Background] Feld R, Woodside DB, Kaplan AS, Olmsted MP, Carter JC. Pretreatment motivational enhancement therapy for eating disorders: a pilot study. Int J Eat Disord. 2001 May;29(4):393-400. doi: 10.1002/eat.1035. PMID 11285576
- [Background] Casasnovas C, Fernandez-Aranda F, Granero R, Krug I, Jimenez-Murcia S, Bulik CM, Vallejo-Ruiloba J. Motivation to change in eating disorders: clinical and therapeutic implications. Eur Eat Disord Rev. 2007 Nov;15(6):449-56. doi: 10.1002/erv.780. PMID 17960774
- [Background] Carter O, Pannekoek L, Fursland A, Allen KL, Lampard AM, Byrne SM. Increased wait-list time predicts dropout from outpatient enhanced cognitive behaviour therapy (CBT-E) for eating disorders. Behav Res Ther. 2012 Aug;50(7-8):487-92. doi: 10.1016/j.brat.2012.03.003. Epub 2012 Mar 30. PMID 22659158
- [Background] Austin A, Flynn M, Richards K, Hodsoll J, Duarte TA, Robinson P, Kelly J, Schmidt U. Duration of untreated eating disorder and relationship to outcomes: A systematic review of the literature. Eur Eat Disord Rev. 2021 May;29(3):329-345. doi: 10.1002/erv.2745. Epub 2020 Jun 23. PMID 32578311